CLINICAL TRIAL: NCT06468358
Title: A Phase Ib/II, Open, Dose-escalation and Expansion Study to Evaluate LB1410 in Combination With LB4330 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate LB1410 in Combination With LB4330 in Patients With Advanced or Metastatic Solid Tumors
Acronym: TRIGGERCD8
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: L & L Bio Co., Ltd., Ningbo, China (Industry)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRIGGERCD8
Record Dates: First submitted 2024-05-31; First posted 2024-06-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: This is a Phase Ib/II, open, dose-escalation and expansion study of LB1410 in combination with LB4330 in patients with advanced or metastatic solid tumors. The study includes 2 parts, Part 1 Dose Escalation and Part 2 Dose Expansion. Initially, participants with pancreatic ductal adenocarcinoma, cholangiocarcinoma, colorectal cancer, ovarian, fallopian tube, or primary peritoneal cancer, non-small cell lung cancer, gastric and gastroesophageal junction adenocarcinoma, esophageal squamous cell carcinoma, hepatocellular carcinoma, renal cell carcinoma, cervical squamous cell carcinoma, and endometrial carcinoma will be enrolled in the study; additional tumor types may be explored and added in a future amendment to the CSP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase Ib, Dose Escalation of LB1410 in combination with LB4330 (Experimental): Up to 4 dose cohorts will be enrolled in the dose-escalation part with the standard 3+3 dose escalation algorithm approach.
  Interventions: Drug: LB1410; Drug: LB4330
- Phase II, Expansion Cohorts of LB1410 in combination with LB4330 (Experimental): This part includes IIa and IIb. Phase IIa will be enrolled subjects at the dose level with initial anti-tumor activity observed in Phase Ib, the numbers of patients enrolled in the phase IIa could be adjusted based on previously available safety and preliminary efficacy data; the dose level of the phase IIb is the RP2D dose level determined in the phase Ib. The planned expanded cohorts are as follows:
  Cohort A: pancreatic ductal adenocarcinoma;
  Cohort B: cholangiocarcinoma;
  Cohort C: colorectal cancer;
  Cohort D: recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer;
  Cohort E: other solid tumors (non-small cell lung cancer, gastric or gastroesophageal junction adenocarcinoma, esophageal squamous cell carcinoma, hepatocellular carcinoma, renal cell carcinoma, cervical squamous cell carcinoma, and endometrial carcinoma).
  Interventions: Drug: LB1410; Drug: LB4330

INTERVENTIONS:
Drug: LB1410 — anti-PD-1/TIM3 bispecific antibody
Drug: LB4330 — anti-claudin18.2/IL-10 fusion protein

SUMMARY:
This is a phase Ib/II, open, dose-escalation and expansion study of an anti-PD1/TIM3 bispecific antibody，LB1410 in combination with an anti-Claudin18.2/IL-10 fusion protein, LB4330 in patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The phase Ib/II clinical study in Chinese patients with advanced or metastatic solid tumors to evaluate the safety, pharmacokinetic (PK), pharmacodynamic (PD), anti-tumor efficacy, and biomarkers of LB1410 in combination with LB4330.

The study will include 2 parts: dose escalation (Phase Ib) and dose expansion (Phase II). Repeated intravenous infusion of LB1410 in combination with LB4330 in patients with metastatic or advanced pancreatic ductal adenocarcinoma, cholangiocarcinoma, colorectal cancer, ovarian, fallopian tube, or primary peritoneal cancer, non-small cell lung cancer, gastric and gastroesophageal junction adenocarcinoma, esophageal squamous cell carcinoma, hepatocellular carcinoma, renal cell carcinoma, cervical squamous cell carcinoma, and endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years of age when signing informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 without deterioration in the past 2 weeks.
3. Estimated life expectancy of ≥12 weeks.
4. Baseline IL-6 levels below 40 pg/mL.
5. Histologically or cytologically documented advanced and metastatic solid tumors for which can't tolerate standard treatment, standard treatment fails, or no standard treatment is available at this stage.
6. Must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at screening.
7. Adequate hematologic function prior to registration for protocol therapy defined as the following criteria:

   1. absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, without the use of granulocyte colony-stimulating factor such as filgrastim in the 2 weeks prior to study treatment (≤ 14 days);
   2. platelet count ≥ 120 × 10^9/L, without transfusion or use of drugs like recombinant human platelet growth factor in the 2 weeks prior to study treatment (≤ 14 days), for HCC patients, platelet count ≥ 100 × 10^9/L;
   3. hemoglobin ≥ 90 g/L, without transfusion or use of drugs like erythropoietin in the 2 weeks prior to study treatment (≤ 14 days).
8. Both AST and ALT ≤ 3 × ULN (both AST and ALT < 5 × ULN for subjects with known hepatocellular carcinoma or hepatic metastases); total bilirubin ≤ 1.5 × ULN (except for subjects with elevated serum bilirubin due to documented underlying conditions such as Gilbert's syndrome or familial benign unconjugated hyperbilirubinemia); for bile duct cancer patients, total bilirubin ≤ 2 × ULN; and serum albumin ≥ 30 g/L.
9. Adequate renal function defined as: serum creatinine ≤ 1.5 × ULN, and creatinine clearance ≥ 50 mL/min (calculated by Cockcroft-Gault formula).
10. Requirements for coagulation function are as follows:

    1. activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN;
    2. international normalized ratio (INR) ≤ 1.5 × ULN (INR ≤ 3 × ULN for subjects receiving warfarin anticoagulant therapy).
11. Any prior anti-tumor therapies (including endocrine/chemotherapy/targeted therapy/immunotherapy) before treatment should washout:

    1. at least 4 weeks for biological therapy (e.g., antibodies);
    2. at least 2 weeks or 5 half-lives (whichever is longer) for small molecule drugs, including 5-FU or its derivatives; at least 6 weeks for nitrosoureas and mitomycin;
    3. at least 2 weeks for Chinese herbal medicine used for indications of anti-tumor activity;
    4. at least 4 weeks for any systemic therapeutic investigational drugs;
    5. at least 2 weeks for any radiotherapy;
    6. any related toxicities or prior adverse events resolved to baseline or ≤ NCI CTCAE 5.0 grade 1 (excluding toxicities without safety risk judged by the investigator, such as alopecia, grade 2 peripheral neuropathy, stable hypothyroidism under hormone replacement therapy, etc.).
12. Phase Ib dose escalation additional inclusion criteria: histologically or cytologically documented advanced malignant solid tumors (preferably pancreatic ductal adenocarcinoma, cholangiocarcinoma, ovarian cancer, microsatellite stable colorectal cancer, advanced solid tumors previously treated with anti-PD-1/PD-L1 inhibitors, such as gastric or gastroesophageal junction adenocarcinoma, or other solid tumors determined by the investigator and sponsor);
13. Phase II (phase IIa and IIb) dose expansion cohort A additional inclusion criteria:

    1. must have received at least one but no more than two prior lines of systemic therapy;
    2. CA199 < 1000 IU/mL during screening period
    3. must not have received any immune checkpoint inhibitor (ICI) therapy.
14. Phase II (phase IIa and IIb) dose expansion cohort B additional inclusion criteria:

    1. must have received at least one but no more than three prior lines of systemic therapy;
    2. without C-Met, FGFR, IDH1 mutations or the genotype is unknown;
    3. CA199 < 1000 IU/mL during screening period.
15. Phase II (phase IIa and IIb) dose expansion cohort C additional inclusion criteria:

    1. must have received at least one but no more than three prior lines of systemic therapy;
    2. CA199 < 1000 IU/mL during screening period;
    3. must not have received any immune checkpoint inhibitor (ICI) therapy;
    4. KRAS, NRAS and BRAF are wild type;
    5. without hepatic metastasis.
16. Phase II (phase IIa and IIb) dose expansion cohort D additional inclusion criteria:

    1. recurrent epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer;
    2. must have received at least one but no more than three prior lines of systemic therapy;
    3. must not have received any immune checkpoint inhibitor (ICI) therapy;
    4. PD-L1 positive;
    5. have received one prior treatment regime of platinum-based chemotherapy;
    6. subjects with BRCA germline mutation (gBRCA mut) should been treated with a polyADP ribose polymerase inhibitor (PARPi), such as Olaparib, Rucaparib, or Niraparib.
17. Phase II (phase IIa and IIb) dose expansion cohort E additional inclusion criteria:

    1. includes non-small cell lung cancer, gastric or gastroesophageal junction adenocarcinoma, esophageal squamous cell carcinoma, hepatocellular carcinoma, kidney carcinoma, cervical squamous cell carcinoma, and endometrial carcinoma;
    2. must have received at least one but no more than two prior lines of systemic therapy, of which only one prior line of therapy contained an anti-PD-1/PD-L1;
    3. subjects with PD-1/PD-L1 primary resistance are required to be known PD-L1 positive.

       For NSCLC,
       1. non-squamous NSCLC must have documented test results of EGFR mutation, ALK fusion and ROS1 fusions, and the above driver genes must be wild type;
       2. non-squamous NSCLC, if RET, MET, NTRK gene testing has been performed previously, the results must be wild type;
       3. squamous NSCLC, if EGFR, ALK fusion gene and ROS1 fusion gene testing has been performed previously, the results must be wild type.

       For ESCC,
       1. exclude a history of gastrointestinal perforation and/or fistula within 6 months prior to initial medication;
       2. after esophageal or tracheal stent implantation is excluded.

       For HCC
       1. Barcelona Clinic Liver Cancer (BCLC) stage C and stage B;
       2. liver function status Child-Pugh (CP) class A and class B in good status(≤7 points);
       3. exclude: a) known fibrolamellar HCC, sarcomatiod HCC, intrahepatic cholangiocarcinoma, or mixed hepatocellular carcinoma and cholangiocarcinoma and other histological types; b) tumor thrombus intrudes into the main and branches of large blood vessels such as portal vein, superior mesenteric vein or inferior vena cava, and causes complications such as portal hypertension and jaundice, or has related clinical risks judged by the researchers to be unsuitable for participation in this study; c) local to regional treatment for the liver (i.e., transarterial chemoembolization, transcatheter embolization, hepatic arterial infusion, radiotherapy, radioembolization, or ablation) within 4 weeks prior to initial medication.

       For RCC Clear cell renal cell carcinoma with or without sarcomatoid components.

       For EC
       1. histopathology confirmed Stage III/IV epithelial endometrial carcinoma including endometrioid carcinoma, non-endometrioid carcinoma, and carcinosarcoma;
       2. non-known ER, PR positive endometrial cancer.

       Note: neoadjuvant ± adjuvant therapy is considered as one of treatment line; maintenance treatment as part of the former first-line treatment.

       PD-L1 positive is defined as PDL1 TPS≥1%, IPS≥1% or CPS≥1.
18. Non-pregnant women and willingness of female participants to avoid pregnancy or male participants willing to avoid fathering children through highly effective methods of contraception after signing informed consent, during the study period, and within 6 months after the last medication.
19. Fully understand the informed consent and sign voluntarily.
20. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

exclusion criteria:

1. Pregnancy, lactation, or breastfeeding.
2. Any prior ≥ Grade 3 immune-related adverse events (irAEs) while receiving immunotherapy or any grade irAE leading to discontinuation in prior immunotherapy; or grade 4 myelosuppression during prior antitumor therapy.
3. Known history of allergy or severe hypersensitivity reactions to other monoclonal antibodies or intravenous immunoglobulins such as anti-PD1/anti-PD-L1 antibodies, TIM-3, interleukin-10, or any of its excipients.
4. Active autoimmune disease or symptomatic history of autoimmune disease (including celiac disease) requiring pharmacological doses of systemic corticosteroids and/or immunosuppressive. Exceptions include vitiligo, relieved asthma/atopic disease, type 1 diabetes or hypothyroidism treatable with alternative therapy and achieving clinical stability during screening, or any other autoimmune disease after discussion with the principal investigator and sponsor.
5. Requirement for systemic corticosteroids (≥ 10 mg/day prednisone or equivalent) or other immunosuppressive therapy within 14 days prior to the planned first dose of study intervention. Inhalational or topical corticosteroids and adrenal replacement steroids (≤ 15 mg prednisone once daily equivalent) are allowed in the non-active autoimmune disease. Ophthalmic, nasal, inhaled, and intra-articular corticosteroids are allowed; short-term use of glucocorticoids for prophylactic treatment (e.g., prevention of contrast media allergy) is allowed.
6. Any of the following prior treatments:

   1. major surgical procedure (e.g., laparotomy, thoracotomy, organ resection, etc.), severe trauma, etc. (Replacement of intravenous drip droppers is acceptable) within 4 weeks prior to first dose, or not recovered from prior surgery; surgery within 14 days prior to the first dose to improves tumor complications or reduces tumor risk (e.g., cervical cancer subjects undergoing nephrostomy or urethral stent placement); significant surgery planned within 30 days after the first dose (except for local surgeries such as placement of systemic ports, core needle biopsy, and prostate biopsy, provided the surgery is completed at least 24 hours before the first dose of study intervention);
   2. receipt of live vaccine or live attenuated vaccine within 4 weeks prior to first dose of study intervention;
   3. use of modulating drugs within 14 days prior to first dose of study intervention, including but not limited to thymosin peptide, interleukin-2, interferon, etc.;
   4. history of allogeneic organ transplant, allogeneic hematopoietic stem cell transplant, or bone marrow transplant.
7. Prior use of drugs with the same mechanism of action as the study drug (e.g., anti-PD1 antibody in combination with anti-TIM3 antibody, PD1/TIM3 bispecific antibody, or IL-10-containing drug).
8. Active infection including syphilis, hepatitis B (HBsAg positive and HBV-DNA > 200 IU/mL or 1000 cps/mL or HBV DNA above the lower limit of detection if the lower limit of the study center is above 200 IU/mL), hepatitis C (Patients with HCV antibody positive but HCV-RNA < lower limit of the study center were admitted).
9. History of other malignant tumors within the past 3 years.
10. Subjects with meningeal metastasis, spinal cord compression, or symptomatic unstable brain metastases or requiring steroids and/or antiepileptic drugs within 4 weeks before enrollment.
11. Severe infection requiring systemic antibiotic therapy within 14 days prior to first dose, or active infection requiring systemic treatment.
12. Uncontrolled or poorly controlled diabetes (glycated hemoglobin ≥ 7.5 at screening), asthma, chronic obstructive pulmonary disease, or other diseases that pose a risk to study participants.
13. Any syncope or seizure within 28 days prior to first dose of the study intervention.
14. Known gastric bleeding lesions or patients considered to be at high risk of gastric bleeding by the investigator.
15. Known presence of diseases such as symptomatic irritable bowel syndrome (such as chronic nausea, persistent recurrent vomiting or diarrhea) and gastric bleeding or intestinal obstruction.
16. Known history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    1. uncontrolled cardiovascular diseases within 3 months before the study, including but not limited to congestive heart failure required treatment (NYHA > II), uncontrolled hypertension (resting blood pressure ≥ 160/100 mmHg), uncontrolled arrhythmia;
    2. myocardial infarction, unstable angina, viral myocarditis, pericarditis, cerebrovascular accident, or other acute uncontrolled heart disease within the recent 6 months;
    3. Electrocardiogram: Female QTcF > 470 milliseconds (ms), Male QTcF > 450 ms (QTcF = QT/RR1/3), or congenital long QT syndrome;
    4. Echocardiographic assessment: Left ventricular ejection fraction (LVEF) ≤ 50% measured by multiple-gated acquisition (MUGA) or echocardiography.
17. Known evidence of interstitial lung disease, symptomatic or may interfere with suspicious findings or management of drug-related pulmonary toxicity.
18. Active tuberculosis (TB).
19. Positive human immunodeficiency virus (HIV).
20. Diseases involving the central nervous system (except for patients with prior brain metastases treated at least 4 weeks before first dose, clinically stable, and not requiring long-term corticosteroid therapy) or history of NCI CTCAE 5.0 Grade 3 or higher drug-related central nervous system toxicity.
21. Venous/arterial thrombotic events occurred within 6 months, including cerebrovascular accidents (such as transient ischemic attacks, cerebral hemorrhage, cerebral infarction such as lacunar infarcts), deep venous thrombosis, and pulmonary embolism.
22. Uncontrolled pleural effusion, pericardial effusion, or ascites (clinically significant recurrence requiring additional intervention every 2 weeks or more frequently).
23. History of severe psychiatric disorders, substance abuse, alcoholism, or drug abuse.
24. Have experienced ≥ grade 3 infusion-related reactions to protein therapeutics.
25. Any other disease (including severe medical or psychiatric conditions) or significant clinical laboratory abnormalities judged by the investigator to potentially affect subject safety, study integrity, or subject's willing in the study.
26. All known MSI-H/dMMR patients.
27. All known HER-2 positive (IHC 3+ or IHC 2+, Fish amplification) patients.
28. Urine protein ≥ 2+, and 24-hour urine protein quantification ≥ 1.0g.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability (Adverse Event reported per NCI-CTCAE v5.0) | up to 60 days following last dose
  Incidence of treatment-emergent adverse events (TEAEs) and treatment-related adverse events reported per NCI-CTCAE v5.0
Incidence and severity of serious adverse events (SAEs) and other special interest (immune-related AEs) | up to 60 days following last dose
  According to NCI-CTCAE v5.0
Incidence of Dose limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  The DLT for this study is defined per CTCAE 5.0 and will be evaluated in the Cycle 1 of treatment in the dose escalation part. If dosing delay occurs, the DLT evaluation should be correspondingly extended to 14 days after the second dosing.
Maximum tolerance toxicity (MTD) and recommended dose for Phase II (RP2D) definition | up to 1 year
  MTD and RP2D based on the safety data collected during the dose escalation phase (Phase I)
Overall response rate (ORR) | From first participant until last participant assessment, an average of 8 months
  Percentage of patients whose best overall response is either a Complete Response or a Partial Response according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) criteria over the total number of evaluable patients
Disease control rate (DCR) | From first participant until last participant assessment, an average of 8 months
  Percentage of patients whose best overall response is either a Complete Response, a Partial Response or Stable Disease according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) criteria over the total number of evaluable patients.
Duration of overall Response (DoR) by RECIST version 1.1 | From first participant until last participant assessment, an average of 8 months
  Time from the date of first documented response (CR or PR) to the date of first documented disease progression according to RECIST 1.1 criteria or the date of death due to underlying cancer.
Progression Free Survival (PFS) by RECIST version 1.1 | From first participant until last participant assessment, an average of 8 months
  Time from the first infusion of LB1410 and LB4330 to the date of first documented tumor progression according to RECIST 1.1 criteria or death due to any cause, whichever occurs first over evaluable patients.
DDC | From first participant until last participant assessment, an average of 8 months
  Time from the date of first documented CR, PR or SD to the date of first documented disease progression according to RECIST 1.1 criteria or the date of death due to any cause.
Overall Survival (OS) duration | From first participant until last participant assessment, an average of 1 year
  Time from first LB1410 and LB4330 infusion to the date of death due to any cause over evaluable patients.

SECONDARY OUTCOMES:
Pharmacokinetics of LB1410 and LB4330: Maximum plasma concentration of the study drug (Cmax) | Through study completion, an average of 1 year
  Maximum observed plasma concentration of the study drug
Pharmacokinetics of LB1410 and LB4330: Area Under the concentration-time curve (AUC) | Through study completion, an average of 1 year
  Area under the plasma concentration-time curve
Pharmacokinetics of LB1410 and LB4330: Clearance | Through study completion, an average of 1 year
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time
Pharmacokinetics of LB1410 and LB4330: Terminal elimination half-life ( T½) | Through study completion, an average of 1 year
  Terminal elimination half life
Evaluation of immunogenicity of each antibody drug in the combinations | Up to 60 days following last dose
  Occurrence of anti-drug antibody (ADA) measured in serum at selected time points during the study

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China